CLINICAL TRIAL: NCT02288182
Title: A Randomized Controlled Clinical Trial to Investigate the Capability of Straumann® VivOss™ Compared to Geistlich Bio-Oss® in Sinus Floor Augmentation
Brief Title: Randomized, Controlled Study to Compare Straumann® VivOss™ to Geistlich Bio-Oss® in Sinus Floor Augmentation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR03/13
Record Dates: First submitted 2014-10-28; First posted 2014-11-11 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Healthy
Keywords: Sinus augmentation procedure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Straumann VivOss (Experimental): Straumann® VivOss™Straumann® VivOss™, is a synthetic bone graft substitute in granulated form. It consists of > 90% TCP (Tri-Calcium-Phosphate -Ca3(PO4)2) and < 10% Hydroxyapatite (Ca10(PO4)6 (OH)2). The granules have a size of 250-1000 μm.
  Interventions: Device: Straumann VivOss
- Geistlich Bio-Oss (Active Comparator): The control device is Geistlich Bio-Oss® spongiosa granules (Geistlich Pharma AG, Wolhusen, Switzerland), 0.25-1 mm in diameter. It's a natural bone mineral of bovine origin. It shall be used according to the instructions of the manufacturer.
  Interventions: Device: Geistlich Bio-Oss

INTERVENTIONS:
Device: Straumann VivOss — Patients will receive Straumann VivOss for sinus augmentation.
  Arms: Straumann VivOss
Device: Geistlich Bio-Oss — Patients will receive Geistlich Bio-Oss for sinus augmentation.
  Arms: Geistlich Bio-Oss

SUMMARY:
A randomized controlled clinical trial to investigate the capability of Straumann® VivOss™ compared to Geistlich Bio-Oss in sinus floor augmentation to demonstrate superiority of Straumann® VivOss™ compared to Geistlich Bio-Oss in regards to the ratio of newly formed bone to residual bone substitute.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled study. The total study duration for each patient should be 9-14 months (from screening to last visit).

Enrolled subjects are randomized to one of the following groups:

1. Sinus floor elevation with Straumann® VivOss™
2. Sinus floor elevation with Geistlich Bio-Oss®

In total 6 visits per patient are scheduled in this study. The histological evaluation of the ratio of newly formed bone to residual bone graft, survival and success rate of study implants and adverse events (AEs) will be assessed.

The study devices Straumann® VivOss™ and Geistlich Bio-Oss are CE-(Conformité Européenne, meaning European Conformity) marked products.

Two centers, one in Germany and one in Switzerland will participate.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have voluntarily signed the informed consent before any study related action
* Males and females with at least 18 years of age (including 18 years)
* Subject needs augmentation procedure in the sinus to prepare for implant placement.
* Subject must have a residual bone height of 2 to 4 mm.
* Adequate oral hygiene ((Full mouth plaque index (O'Leary, et al. 1972 ) <25%) at baseline
* Adequate control of inflammation ((full mouth bleeding on probing (Ainamo and Bay 1975)) ≤25% at baseline

Exclusion Criteria:

* Systemic disease that would interfere with bone or wound healing and dental implant therapy (e.g. uncontrolled diabetes)
* Systemic disease that would interfere with bone or wound healing and dental implant therapy (e.g. uncontrolled diabetes)
* Any contraindications for general bone grafting and oral surgical procedures
* Any anomalies of the sinus that could interfere with planned procedures
* History of local irradiation therapy
* Local inflammation, including untreated periodontitis
* Medical conditions requiring chronic high dose steroid therapy
* Treatment with an investigational drug or device within a 30 day period immediately prior to surgery at visit 2, or expected participation in any other investigational drug or device study during the conduct of this trial.
* Antibiotic treatment or anti-inflammatory treatment within 4 weeks prior to surgery
* History of alcoholism or drug abuse
* Immunocompromised subjects
* Subjects who smoke >10 cigarettes per day or tobacco equivalents or chew tobacco
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance or unreliability
* Physical or mental disabilities that would interfere with the ability to perform adequate oral hygiene
* Current pregnancy (pregnancy test) and breastfeeding women

Secondary exclusion criterium:

Defects of the Schneider Membrane

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Jung, PD, Principal Investigator — University of Zurich
Locations (2):
- Zentrum für Implantologie, Parodontologie und 3D- Diagnostik, Konstanz, Baden-Wurttemberg, Germany
- University of Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buser D, Weber HP, Lang NP. Tissue integration of non-submerged implants. 1-year results of a prospective study with 100 ITI hollow-cylinder and hollow-screw implants. Clin Oral Implants Res. 1990 Dec;1(1):33-40. doi: 10.1034/j.1600-0501.1990.010105.x. PMID 2099210

RESULTS

PARTICIPANT FLOW:
Groups:
- Straumann VivOss; Geistlich Bio-Oss: Subjects were randomized either to the test group receiving Straumann VivOss oder comparator group receiving Geistlich Bio-Oss. If a patient needed augmentation in both sinuses, one sinus was randomized into the test group receiving Straumann VivOss and the other (opposite) sinus should be treated with Geistlich Bio-Oss. In those bilateral patients, biopsies were taken from both sinuses.
Period: Overall Study
Arm/Group | Straumann VivOss | Geistlich Bio-Oss
Started | 25 | 27
Completed | 25 | 25
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT Data Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Straumann VivOss | Geistlich Bio-Oss | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (11.8) | 60.3 (9.9) | 59.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 7 | 10 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 24 | 25 | 49
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Newly Formed Bone to Residual Bone Graft in Patients Treated With Straumann® VivOss™ Compared to Geistlich Bio-Oss®
Description: Bone biopsies and histological staining
Time Frame: 6 months +/- 7 days after bone augmentation
Population: The biopsies were retrieved from the central part of the dental implant osteotomy. In patients with bilateral treatment, biopsies were taken from both sinuses.
Measure: Median (Inter-Quartile Range); unit: ratio
Units Other Than Participants: biopsies
Groups:
- Straumann VivOss: Straumann® VivOss™, is a synthetic bone graft substitute in granulated form. It consists of > 90% TCP (Tri-Calcium-Phosphate -Ca3(PO4)2) and < 10% Hydroxyapatite (Ca10(PO4)6 (OH)2). The granules have a size of 250-1000 μm.
  Straumann VivOss: Patients will receive Straumann VivOss for sinus augmentation.
Arm/Group | Straumann VivOss | Geistlich Bio-Oss
Number analyzed (Participants) | 25 | 25
Number analyzed (biopsies) | 29 | 33
ratio | 1.37 [1.00 to 2.22] | 0.69 [0.58 to 1.05]
Statistical Analysis 1: Comparison: Straumann VivOss vs Geistlich Bio-Oss; Student's t-test comparing the group means was planned and performed (successfully). However, due to some outliers, the central tendencies have been reported as medians (instead of arithmetic means). Therefore an additional non-parameteric test (Mann-Whitney U-test) was performed; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Survival Rate of Study Implants (Based on Subjects)
Description: Number of implants in place
Time Frame: 4 months +/- 1 month after implant placement
Population: ITT Data Set
Measure: Count of Participants; unit: Participants
Arm/Group | Straumann VivOss | Geistlich Bio-Oss
Number analyzed (Participants) | 25 | 25
Participants | 24 | 22

3. Secondary Outcome: Success Rate of Study Implants
Description: Buser success criteria:
  * Absence of persisting subjective discomfort such as pain, foreign body perception and or dysaesthesia (painful sensation)
  * Absence of a recurrent peri-implant infection with suppuration (where an infection is termed recurrent if it is observed at two or more follow-up visits after treatment with systemic antibiotics)
  * Absence of implant mobility on manual palpation
  * Absence of any continuous peri-implant radiolucency.
Time Frame: 4 months +/- 1 month after implant placement
Population: ITT Data Set
Measure: Count of Participants; unit: Participants
Arm/Group | Straumann VivOss | Geistlich Bio-Oss
Number analyzed (Participants) | 25 | 25
Participants | 25 | 25

4. Other Pre Specified Outcome: Basic Bone Situation
Description: This measure describes the basic bone situation of the patients at baseline, i.e. the bone thickness as a unit of area before the application of bone substitute material.
Time Frame: 6 months +/- 7 days after bone augmentation
Population: ITT Data Set
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Straumann VivOss | Geistlich Bio-Oss
Number analyzed (Participants) | 25 | 25
mm^2 | 1.50 (0.42) | 1.27 (0.43)

ADVERSE EVENTS:
Time Frame: Overall study period (10 months per patient)
Arm/Group | Straumann VivOss | Geistlich Bio-Oss
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/27
Other Adverse Events (participants affected / at risk) | 7/25 | 6/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Straumann VivOss (N=25) | Geistlich Bio-Oss (N=27)
urinary tract infection (leading to hospitalization) (Renal and urinary disorders) | 0 (0) | 1 (1) — This was an unexpected event withount any causal relationship to study procedures or devices.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Straumann VivOss (N=25) | Geistlich Bio-Oss (N=27)
implant loss (Product Issues) | 0 (0) | 3 (4)
swelling (General disorders) | 2 (2) | 1 (1)
pain (General disorders) | 2 (2) | 0 (0)
injury (General disorders) | 1 (1) | 0 (0)
compromised wound healing (General disorders) | 1 (1) | 0 (0)
dehiscence (General disorders) | 0 (0) | 1 (1)
explantation (Product Issues) | 1 (1) | 0 (0)
infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT02288182/Prot_SAP_000.pdf